CLINICAL TRIAL: NCT05864157
Title: Targeted Motor Learning to Improve Gait for Individuals With Parkinson Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0021; R21HD111833 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: Gait; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Participants will perform walking practice on a treadmill and overground without the use of a metronome.
  Interventions: Other: Gait training without rhythmic auditory cues
- Targeted Rhythmic Auditory Cueing (TRAC) (Experimental): Participants will perform walking practice on a treadmill (with a metronome set to 85% of typical cadence) and overground (with a metronome set to 115% of typical cadence).
  Interventions: Other: TRAC
- Distorted Targeted Rhythmic Auditory Cueing (dTRAC) (Experimental): Participants will perform walking practice on a treadmill (with a metronome set around 85% of typical cadence) and overground (with a metronome set around 115% of typical cadence).
  Interventions: Other: dTRAC

INTERVENTIONS:
Other: Gait training without rhythmic auditory cues — Gait training on treadmill and overground without any rhythmic auditory cues
  Arms: Control
Other: TRAC — Metronome set to 85% on treadmill and 115% when walking overground
  Arms: Targeted Rhythmic Auditory Cueing (TRAC)
Other: dTRAC — Metronome set around 85% on treadmill and around 115% when walking overground
  Arms: Distorted Targeted Rhythmic Auditory Cueing (dTRAC)

SUMMARY:
The purpose of this research study is to determine how training to step with a metronome on both a treadmill, as well as overground, will influence the way that people with Parkinson disease walk. Using metronomes is commonly used in clinics, but the investigators will be using a combination of slow and fast frequencies to alter the way that people walk. The use of a slower frequency metronome on the treadmill is intended to help participants take larger steps. The use of a faster frequency metronome while walking overground is intended to help participants take faster steps.This will take place over 12 training sessions. Each session will be about an hour. It will include some walking tests and pictures of the brain (using MRI) before and after training.

DETAILED DESCRIPTION:
Some details regarding the metronome frequency are purposely omitted at this time to preserve scientific integrity. They will be included after the trial is complete

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's disease (Hoehn and Yahr Stage 2-3)
* self-report the ability to walk uninterrupted for 10 minutes both overground and on a treadmill without therapist assistance
* comfortable gait speed > 0.4 m/s and < 1.2 m/s
* normal (or corrected to normal [i.e., hearing aid]) hearing
* deficits in gait continuity (e.g., shuffling, shortened strides, freezing, festination, bradykinesia, etc) based on observational gait analysis
* Movement Disorders Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS-III) item 10 ≥1 and <3
* be on stable doses of orally-administered levodopa
* age 50-80 years old

Exclusion Criteria:

* contraindications to MRI (e.g., metal implants, claustrophobia, etc)
* cognitive deficits (Montreal Cognitive Assessment [MoCA] < 26)
* concurrent Physical Therapy
* have undergone deep brain stimulation surgery
* cannot walk without therapist assistance
* uncontrolled cardiorespiratory/metabolic disease, or other neurological disorders or orthopedic injury that may affect gait.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Change in Six minute walk test (6MWT) at the 3 month follow up visit | Baseline, 3 month follow-up
  The 6-minute walk test provides a more objective quantitative measure of mobility, functional performance, and symptom control. It measures the distance an individual can walk over a total of six minutes on a hard, flat surface. The individual can self-pace and rest as needed as they walk back and forth along a marked course. The participant can use an assistive walking device they normally use, such as a cane. The minimum clinically important difference in 6-minute walk distance is approximately 30 meters, a difference that is associated with mortality. A higher change score represents a greater improvement in walking function and a better outcome.

SECONDARY OUTCOMES:
Change in Six minute walk test (6MWT) after 4 weeks of training | baseline, 4 weeks
  The 6-minute walk test provides a more objective quantitative measure of mobility, functional performance, and symptom control. It measures the distance an individual can walk over a total of six minutes on a hard, flat surface. The individual can self-pace and rest as needed as they walk back and forth along a marked course. The participant can use an assistive walking device they normally use, such as a cane. The minimum clinically important difference in 6-minute walk distance is approximately 30 meters, a difference that is associated with mortality. A higher change score represents a greater improvement in walking function and a better outcome.
Walking stride length | up to 3 month follow-up
  The walking stride length represents the average stride length (distance between where one foot strikes the ground to the location that the same foot strikes the ground to complete the stride). The distance is measured from walking over a pressure mat during the 6MWT. This measurement will be completed at baseline (prior to training), after 4 weeks of training, and again for a 3 month follow-up. A larger value represents longer steps, and a better outcome.
Walking Cadence | up to 3 month follow-up
  Walking cadence is the frequency of steps per minute (inverse of step time). The average cadence is measured from passes over a pressure mat during the 6MWT, and will be completed at baseline (prior to training), after 4 weeks of training, and again for a 3 month follow-up.
Gait interruption index | up to 3 month follow-up
  The Gait Interruption Index represents the number of 'freezes' observed, divided by the number of 'freeze opportunities' (i.e., turns, times stepping on/off pressure mat) completed during the 6MWT. A higher number represents greater impairment in Freezing of Gait. This measurement will be completed at baseline (prior to training), after 4 weeks of training, and again for a 3 month follow-up.
Mini BESTest (Balance Evaluation Systems Test) score | up to 3 month follow-up
  The mini-BESTest is a 14-item, clinical battery used to assess balance in four component areas (anticipatory transitions, postural response, sensory orientation and dynamic gait) and provides a single number summary of balance performance. Scores range from 0 to 28 with higher scores indicate higher function.
Freezing of Gait Questionnaire score | up to 3 month follow-up
  The Freezing of Gait Questionnaire assesses freezing of gait (FOG) severity unrelated to falls in patients with Parkinson disease (PD), FOG frequency, disturbances in gait, and relationship to clinical features conceptually associated with gait and motor aspects. The total score ranges from 0-24, with higher scores representing greater severity of FOG symptoms.
Hippocampal volume | up to 4 weeks
  Hippocampal volume represents the size of the hippocampus, which is a portion of the deep brain. In particular, the investigators will compute the three dimensional volume of the hippocampus from structural MRI (Magnetic Resonance Imaging) taken at baseline and after 4 weeks of training.
Fractional anisotropy | up to 4 weeks
  Fractional anisotropy (FA) is derived from diffusion tensor imaging (DTI) sequences taken during the neuroimaging testing. FA reflects a ratio of the directional flows of water molecules within axonal bundles.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Lewek, PT, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected will be shared with other researchers. Specifically, the investigators will share all individual level 6MWT distances, average cadence, stride length, and gait interruption indices from the baseline test, after 4 weeks of training, and at the 3 month follow-up. All MiniBESTtest total scores, and FOGQ total scores from these timepoints will also be shared for each individual. Finally, the investigators will share hippocampal volume and fractional anisotropy values from each participant taken at baseline and after four weeks of training.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Moreover, the investigators are committed to releasing all data, including neuroimaging, and scale data to the general scientific community, upon completion of the study. In particular, the investigators will use open platforms (e.g., UNC Dataverse) to disseminate data. Access to the data repository will be free of charge.